CLINICAL TRIAL: NCT01895673
Title: The Use of PET-MRI in the Follow-up of RFA and MWA Treated Colorectal Liver Metastases
Brief Title: PET-MRI After Radiofrequency Ablation (RFA) or Microwave Ablation (MWA)
Status: Completed | Type: Observational
Sponsor: dr. M.P. van den Tol MD PhD (Other)
Responsible Party: Sponsor-Investigator, dr. M.P. van den Tol MD PhD, PhD, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Other Study IDs: NL43058.000.13
Record Dates: First submitted 2013-06-20; First posted 2013-07-10 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Liver Neoplasms; Local Neoplasm Recurrence
Keywords: FDG-PET; Radiofrequency Ablation; Magnetic Resonance Imaging
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Recurrence, Local | interventions — Gadolinium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PET-MRI: Twenty patients with RFA/MWA for CRLM or RFA/MWA of recurrent liver lesions after prior local treatment of CRLM and are eligible to undergo MRI-scanning are included when they have adequate renal function. Patients that do not meet inclusion criteria for undergoing an MRI scan are excluded.
  Interventions: Other: Gadolinium

INTERVENTIONS:
Other: Gadolinium — All patients will undergo PET-MRI additional to the PET-CT they routinely undergo. All patients will be administered Gadolinium for the PET-MRI scan. This is an extra intervention than they would normally undergo.

SUMMARY:
The primary objective of this study is to evaluate the ability of PET-MRI and to detect a local site recurrence during the first year of follow-up after RFA or MWA of colorectal liver metastases (CRLM) as compared with contrast enhanced (ce) CT and PET-CT. Standard reference will be clear focal uptake in the rim of the lesion on PET-CT, possibly in combination with histology (when available) or clinical follow-up.

Secondary outcomes are the inter-observer variability, the ability to diagnose new intrahepatic lesions and in what way PET-MRI is able to influence future treatment compared to PET-CT and ceCT. The patients satisfaction concerning the PET-MRI will be examined with a questionnaire.

DETAILED DESCRIPTION:
All included patients will routinely undergo follow-up with 3 monthly ceCT of the liver and PET-CT in the first year after RFA/MWA of CRLM according to standard of care in our hospital. Patients are asked to undergo an additional PET-MRI of the liver on the same day in the first year (in total 4 scans). The PET-MRI is obtained before the PET-CT. The 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) used for PET-CT and PET-MRI are alike and one injection is sufficient. The PET-CT has to be made within 150 minutes after FDG injection. Anonymous PET-MRI results are independently reviewed by 2 experienced radiologists and 2 nuclear medicine physicians twice, with a time-interval of at least two weeks between the first and second review. Based on these results, treatment decisions will be compared for any change in decision making.

The evaluate inter-observer variability we will ask the two nuclear medicine physicians and two radiologist to assess all results and score local and intrahepatic tumor progression. Results of the first and second evaluation will be compared to determine inter observer agreement using Cohen's Kappa. Local recurrence and new lesions will be scored on a separate form with standard criteria.

The reports on LSR will be scored as follows:

* Normal: when the reviewer is sure that no tumor recurrence is present in the ablation zone.
* Probably benign: FDG is enhanced, but compatible with post-ablation inflammation or rim-like characteristics on MRI images (not focal!)
* Equivocal: there is doubt whether the enhanced FDG, CT- or MRI features are due to tumor recurrence or inflammation
* Probably malign: when the reviewer is sure about local recurrence in the ablation zone. Size and location will also be reported.

The reports on new intrahepatic lesions will be scored as follows:

* Normal: no new intrahepatic disease outside 1cm of the ablation zone
* Equivocal: doubt about the malignant origin of a lesion
* Probably malign: new intrahepatic tumor not within 1cm of the ablation zone, including size and location.

The results of all scans by the reviewers, in the way as described above, will be compared to each other to determine the inter-observer variability using Cohen's Kappa.

A questionnaire with 7 questions is completed at the end of one year follow-up to determine patients experience with PET-MRI and PET-CT.

The questions will be in Dutch, but are translated below for this purpose. Patients can answer on a scale 1-5 and n/a.

* The PET-MRI was less burdensome than PET-CT
* The PET-MRI was more bothersome than I expected
* PET-MRI is more comfortable than PET-CT
* If I could choose, I would rather undergo PET-MRI than PET-CT
* The noise of the PET-MRI was annoying
* The fact that PET-MRI takes longer than PET-CT isn't an issue for me
* I would rather undergo a PET-MRI than a PET-CT if results are proven to be equal

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of primary colorectal tumor
* Radiological or histological prove of one or more CRLM or radiological proof of a LSR after previous RFA/MWA treatment for CRLM
* CRLM or LSR treated with RFA/MWA or RFA/MWA in combination with resection
* Follow-up imaging performed in Free University (VU) University Medical Center
* Age ³ 18 years
* Life expectancy of at least 1 year
* estimated glomerular filtration rate (eGFR) > 60 or hydration according to protocol before scanning
* Written informed consent.

Exclusion Criteria:

* cirrhosis or steatosis of the liver
* Chemotherapy ≤ 6 weeks before scanning (during the entire study)
* Pregnant or breast-feeding subjects
* Allergy to contrast media
* Patients developing recurrent intrahepatic disease that require resection of the ablated lesion
* eGFR < 60, unless hydration according to protocol is possible
* General exclusion criteria to undergo MRI

  1. claustrophobia
  2. intracranial clips
  3. any implanted stimulation device (eg. internal cardioverter defibrillator/pacemaker, cochlear implant)
  4. intra-ocular metal splinters or metal clips
  5. Metal artificial heart valve
  6. Bone prosthesis < 6 weeks
  7. inability to lie still for 30 minutes
  8. orthopnea
  9. intestinal video capsule
  10. Metal intra auricular prosthesis

all other prosthesis or piercings should be removed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients with primary CRLM or recurrent liver disease after prior local treatment of CRLM that have been treated with RFA or MWA and are eligible to undergo MRI-scanning are included when they have adequate renal function. Patients that do not meet inclusion criteria for undergoing an MRI scan are excluded.
  Patients are recruted by the study coordinators (K Nielsen or HJ Scheffer) when meeting in- and exclusion criteria from the VU Univeristy medical centre and the Gelderse Vallei hospital in Ede. All scans will be made in the VU University medical centre.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Local site recurrence (LSR) detection | 1 year
  The primary objective of this study is to evaluate the ability of PET-MRI and diffusion and contrast enhanced MRI to detect LSR during the first year of follow-up after RFA treatment of CRLM as compared with ceCT and PET-CT. Standard reference will be clear focal uptake in the rim of the lesion on PET-CT, possibly in combination with histology (when available) or clinical follow-up.

SECONDARY OUTCOMES:
Detection new intrahepatic lesions | 1 year
  the ability of PET-MRI to diagnose smaller new intrahepatic lesions than PET-CT and ceCT
inter-observer variability | 1 year
  Hard copy data sets of all PET-MRI and PET-CT scans, with no patient information, random order, independently reviewed by 2 experienced radiologists and 2 nuclear medicine physicians twice (reviewers blinded to the images and results of the other imaging modalities and blinded to the final outcome of patients), with a time-interval of at least two weeks between the first and second review. These scans are scored on a standardized form (explained in the section 'detailed description'). The outcomes between the different reviewers of the same scan are noted and compared to each other. Inter observer variability is determined using Cohen's Kappa.
Influence on decision making | 1 year
  in what way PET-MRI is able to change future treatment compared to PET-CT and ceCT
Patients experience with PET-CT and PET-MRI | end of one year follow-up
  A questionnaire with 7 questions is completed at the end of one year follow-up to determine patients experience with PET-MRI and PET-CT. This is done to get an idea of the possible objections and wishes of all patients. Results will be described.
  The questions will be in Dutch, but are translated below for this purpose. Patients can answer on a scale 1-5 and n/a.
  * The PET-MRI was less burdensome than PET-CT
  * The PET-MRI was more bothersome than I expected
  * PET-MRI is more comfortable than PET-CT
  * If I could choose, I would rather undergo PET-MRI than PET-CT
  * The noise of the PET-MRI was annoying
  * The fact that PET-MRI takes longer than PET-CT isn't an issue for me
  * I would rather undergo a PET-MRI than a PET-CT if results are proven to be equal

CONTACTS AND LOCATIONS:
Overall Officials: Petrousja van den Tol, MD PhD, Principal Investigator — VU University Medical Centre; Indra C Pieters, MD PhD, Principal Investigator — VU University Medical Centre; Emile FI Comans, MD PhD, Principal Investigator — VU University Medical Centre
Locations (1):
- VU University Medical Centre, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Nielsen K, Scheffer HJ, Pieters IC, van Tilborg AA, van Waesberghe JH, Oprea-Lager DE, Meijerink MR, Kazemier G, Hoekstra OS, Schreurs HW, Sietses C, Meijer S, Comans EF, van den Tol PM. The use of PET-MRI in the follow-up after radiofrequency- and microwave ablation of colorectal liver metastases. BMC Med Imaging. 2014 Aug 8;14:27. doi: 10.1186/1471-2342-14-27. PMID 25103913